CLINICAL TRIAL: NCT04392921
Title: Prophylaxis for Patients at Risk to Eliminate Post-operative Atrial Fibrillation
Acronym: PREP-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20190583-01H
Record Dates: First submitted 2020-05-06; First posted 2020-05-19 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone

STUDY DESIGN:
Intervention Model Description: Prospective, single-centre, double arm pragmatic randomized controlled feasibility trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Patients randomized to amiodarone treatment
  Interventions: Drug: Amiodarone
- Control Arm (Placebo Comparator): Patients randomized to placebo treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amiodarone — Patients will undergo one of the two regimens of amiodarone, based on their ability to tolerate po (per os) intake in the post-operative period:
  • All patient will receive 1050mg of amiodarone in 100mL of 5% dextrose administered intravenously initiated at the time of anesthesia induction at a rate of 0.73mg/min or 43.75mg/h and continued over 24 hours followed by:
  * If able to tolerate po intake: 400mg po BID for post-operative days 1 to 5 or until the day of discharge (whichever occurs first).
  * If unable to tolerate po intake: daily infusion of 1050mg in 100mL of 5% dextrose for postoperative days 1 to 5 or until the day of discharge (whichever occurs first).
  Arms: Intervention Arm
Drug: Placebo — Patients will undergo one of the two schedules or intravenous infusion, based on their ability to tolerate po intake in the post-operative period:
  * All patients will receive 100mL of 5% dextrose administered intravenously initiated at the time of anesthesia induction at a rate of 0.73mg/min or 43.75mg/h and continued over 24 hours followed by:
    o If able to tolerate po intake: 400mg po BID for post-operative days 1 to 5 or until the day of discharge (whichever occurs first).
  * Esophagectomy patient will receive 100mL of 5% dextrose at the time of anesthesia induction at a rate of what would be 0.73mg/min or 43.75mg/h if it contained 1050mg of amiodarone, followed by daily infusion of 100mL of 5% dextrose for 4 days or until the day of discharge (whichever occurs first).
  Arms: Control Arm

SUMMARY:
After surgery on the lungs or esophagus, 12-46% of patients experience an irregular heart rhythm called atrial fibrillation. Although usually transient, post-operative atrial fibrillation is associated with longer stay in hospital, greater complications, and increased risk of death. Several medications have been shown to be effective at reducing the risk of atrial fibrillation after their surgery with the greatest effectiveness and safety demonstrated with amiodarone. Nevertheless, amiodarone has potential side effects, and so it is only recommended in patients with increased risk of developing atrial fibrillation. A tool has been developed and validated to identify high-risk patients but no clinical trial has looked at the effectiveness of administering amiodarone in this high-risk group. This study aims to assess the feasibility and safety of conducting a clinical trial where patients are randomized to receive amiodarone or placebo. This is critical before considering a full-scale trial to assess the effectiveness of amiodarone in reducing atrial fibrillation after surgery on the lungs or esophagus.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or greater
* Undergoing major non-cardiac pulmonary or esophageal surgery (including esophagectomy, pulmonary wedge resection, lobar resection, pneumonectomy, or gastrectomy)
* POAF prediction score greater than or equal to 4

Exclusion Criteria:

* Aged less than 18 years
* History of atrial arrhythmia (paroxysmal or persistent), or Wolf-Parkinson-White syndrome (WPW), or 2nd or 3rd degree heart block without a pacemaker
* Current antiarrythmic therapy (including amiodarone, propafenone, sotalol, flecainide, and dronedarone)
* Previous severe adverse reaction or contraindication to amiodarone (including pre-existing interstitial lung disease, or history of hepatotoxicity from amiodarone)
* QTc interval longer than 450ms
* Serum alanine transaminase or aspartate transaminase over 3 times the upper limit of normal, or Child-Pugh class C
* Allergy to amiodarone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Capability for enrolment | Upon study completion, 1 year following study initiation
  Capacity for enrolment will be assessed, in order to determine recruitment potential and an optimal sample size estimated for a full-scale RCT, by measuring the following outcomes: proportion of patients risk stratified and screened, proportion of eligible individuals consenting to involvement in the study, proportion of recruited individuals who are enrolled in the study.
Proportion of patients randomized who receive the intervention | Upon study completion, 1 year following study initiation
  Feasibility of the randomization process will be evaluated including the proportion of patients randomized who receive the intervention
Knowledge of which patients received intervention and placebo | Upon study completion, 1 year following study initiation
  Feasibility of blinding of participant, care provider, investigator, and outcomes assessor to the intervention allocation of participants will be evaluated by administering a survey to assess their knowledge of which patients received the intervention and placebo
Intervention delivery | Upon study completion, 1 year following study initiation
  Intervention delivery will be assessed by determining if protocol adherence rates exceed >90% and recording observational data on the quality of intervention delivery using a data collection sheet
Protocol compliance | Upon study completion, 1 year following study initiation
  Monitoring of protocol compliance will be measured by the frequency, rate, and rationale of events when study activities diverge from the REB-approved protocol
Adherence to safety protocol | Upon study completion, 1 year following study initiation
  Monitoring of safety will be assessed by determining the rate and efficiency of reporting adverse events if they occur and monitoring adherence rates to safety and monitoring protocols
Proportion of patients for which data could be abstracted | Upon study completion, 1 year following study initiation
  Feasibility of data extraction analysis will be evaluated by the proportion of patients for which the required data could be abstracted: medication use, incidence of post-operative atrial fibrillation, post-operative outcomes, etc.
Resources | Upon study completion, 1 year following study initiation
  Resources required to conduct a future multi-centre PREP-AF trial will be assessed by evaluating the administrative capacity of the POAF research team, including the required number of hours of research assistant time, as well as the feasibility of the designated study budget

SECONDARY OUTCOMES:
Incidence of postoperative atrial fibrillation | Within 30 days post-surgery
  Incidence of postoperative atrial fibrillation, as defined by atrial fibrillation proved by electrocardiogram with an irregular narrow complex tachycardia without p waves
Severity of postoperative atrial fibrillation | Within 30 days post-surgery
  Severity of postoperative atrial fibrillation, as classified by the Clavien-Dindo classification schema, defined for thoracic surgery using the published Ottawa Thoracic Morbidity and Mortality system
Hospital length of stay | Within 30 days post-surgery
  Hospital length of stay, as defined as the number of days inclusive between the day of surgery, and the day of discharge
Other postoperative complications | Within 30 days post-surgery
  Other postoperative complications using the taxonomy of the Ottawa Thoracic Morbidity and Mortality definitions. All complications are recorded with incidence, date, and severity. Of note, post-operative mortality is a grade V complication and is recorded along with its cause as well

CONTACTS AND LOCATIONS:
Overall Officials: Andrew JE Seely, MD, PhD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith HA, Kanji S, Tran DTT, Redpath C, Ferguson D, Lenet T, Sigler G, Gilbert S, Maziak D, Villeneuve P, Sundaresan S, Seely AJE. Prophylaxis for patients at Risk to Eliminate Post-operative Atrial Fibrillation (PREP-AF trial): a protocol for a feasibility randomized controlled study. Trials. 2021 Jun 7;22(1):384. doi: 10.1186/s13063-021-05318-1. PMID 34098992